CLINICAL TRIAL: NCT03947931
Title: Multicenter Prospective Non-randomized Study: Predictors of Colectomy in Patients With Extremely Severe Ulcerative Colitis.
Brief Title: Russian Extremely Severe Ulcerative Colitis Study
Acronym: REXs_UC
Status: Completed | Type: Observational
Sponsor: State Scientific Centre of Coloproctology, Russian Federation (Other Government)
Responsible Party: Principal Investigator, Achkasov Sergey, Achkasov Sergey, Professor of State Scientific Centre of Coloproctology, Head of sugery and oncology of colon department, Moscow, State Scientific Centre of Coloproctology, Russian Federation
Other Study IDs: 127
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Ulcerative Colitis; Inflammatory Bowel Diseases
Keywords: ulcerative colitis, acute severe ulcerative colitis, predictors of colectomy
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General group: Patient with extremely severe ulcerative colitis

SUMMARY:
The purpose of this study is prove the need to selection of a extremely severe ulcerative colitis, to identify predictors of colectomy, which will reduce the optimal time for surgery.

DETAILED DESCRIPTION:
Acute severe ulcerative colitis is a life threatening disease,total mortality rate can reach 17%, and the frequency of surgical treatment approximately 40%. Standard conservative therapy in these patients is often ineffective and the optimal timing of the surgical treatment has not yet been established.

In the Russian clinical guidelines for the treatment of ulcerative colitis, the extremely severe ulcerative colitis is added to the classification of the severity.

The extremely severe ulcerative colitis is a severe, according to the criteria of Truelove, Witts and the endoscopic picture of deep, extensive ulcerative defects of the mucosa, up to the muscular layer with the formation of mucosal islets including albumin reduction.

Conservative treatment of patients with extremely severe ulcerative colitis worsens treatment outcomes only. The authors of the study want to prove that patients with a extremely severe ulcerative colitis need a colectomy in a short time.

Is there a need for long-term follow-up, conservative treatment of high-risk patients? Is it safe to perform early surgical treatment without long-term conservative treatment? This study will allow to answer these questions and help doctors in the treatment of such patients anywhere in Russia and not only.

ELIGIBILITY:
Inclusion Criteria:

* Acute Severe Colitis according to the Truelove and Witt's Criteria;
* Extremely severe activity according endoscopic picture of deep, extensive ulcerative defects of the mucosa, up to the muscular layer with the formation of mucosal islets including albumin reduction (lower 31 g/l).

Exclusion Criteria:

* Pregnancy;
* Infectious, ischemic colitis;
* Transformation of diagnosis into Crohn's disease;
* Medical treatment failure before the admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who admissions with acute severe ulcerative colitis and classified as extremely severe UC.
Sampling Method: Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Inpatient colectomy rate | 30 days
  Operation performed due to the treatment failure and complications during hospitalization.

SECONDARY OUTCOMES:
Long-term colectomy rate | 12 months
Total mortality | 12 months
Postoperative complications | 12 months
  Compared between early and later surgical treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ayrat Mingazov, Study Chair — Sub-investigator
Locations (1):
- State Scientific Centre of Coloproctology, Russian Federation, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No